CLINICAL TRIAL: NCT02192411
Title: Efficacy of Variable Lidocaine Concentrations in Tumescent Anesthesia for Pain Control During and After Endovenous Laser Procedure; a Double Blinded, Randomized, Controlled Non-inferiority Trial
Brief Title: Efficacy of Variable Lidocaine Concentrations in Tumescent Anesthesia for Pain Control During and After Endovenous Laser Procedure; Non-inferiority Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Midwest Vein Center (Other)
Responsible Party: Principal Investigator, Deborah Lindner, MD, Principle Investigator, Midwest Vein Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JVDL070714
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Pain During and After Endovenous Laser Obliteration of Large Saphenous Vein Based on Lidocaine Tumescent Concentration
Keywords: lidocaine; tumescent; endovenous; laser; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Lidocaine (Active Comparator): 50mL 1% lidocaine in 450mL normal saline
  Interventions: Drug: Lidocaine
- 1/4 dose lidocaine (Experimental): 12.5mL 1% lidocaine in 487.5mL normal saline
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — 1/4 dose lidocaine

SUMMARY:
Endovenous laser treatment is a minimally invasive procedure that has been shown to be a safe and effective treatment for varicose veins. Essential to the successful ablation of refluxing veins by endovenous laser treatment is the use of tumescent anesthesia. One of the components of tumescent anesthesia is lidocaine, a commonly used local anesthetic. While lidocaine can be used safely as long as serum concentrations remain low, its use carries the risk of lidocaine toxicity. In order to minimize the risk of lidocaine toxicity it is desirable to use the minimum effective concentration of lidocaine needed to manage pain during a procedure. This study seeks to determine if a ¼ lower concentration of lidocaine in tumescent anesthesia will function as well as the standard dose for pain management in endovenous laser treatments. If we find that this is the case, we will be able to reduce the risk of lidocaine toxicity in patients undergoing endovenous laser treatment, while maintaining their comfort throughout the procedure. This will be achieved through a direct comparison of intra- and post-operative pain for patients randomized to receive either the ¼ tumescent lidocaine concentration or the standard lidocaine concentration.

ELIGIBILITY:
Inclusion Criteria:

* Large Saphenous Vein treatment
* 16-85 years old, good health
* Able to understand informed consent
* Eligible for EVLT determined by physician

Exclusion Criteria:

* Patients with know lidocaine sensitivity
* Bleeding disorders
* Pregnancy
* Congestive heart failure
* Liver dysfunction
* Patient ineligible for EVLT

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Vein Center, Chicago, Illinois, United States